CLINICAL TRIAL: NCT01763359
Title: Decreased Hip Adductor Strength and Obturator Nerve Palsy After the Modified Stoppa Approach to Acetabular Fracture Reduction and Fixation: Is Retraction to Blame?
Brief Title: Hip Strength and Nerve Palsy After the Modified Stoppa Approach to Acetabular Fracture Reduction and Fixation
Status: Terminated | Type: Observational
Why Stopped: The original PI moved on from this facility as did other key personnel. The current PI decided to discontinue the study.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, David Rothberg, M.D., University of Utah
Other Study IDs: 55695
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Acetabular Fracture; Pelvic Fracture
Keywords: acetabular fracture; pelvic fracture; hip adductor strength; obturator nerve palsy; modified Stoppa approach
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this prospective study is to compare hip adductor strength and obturator nerve palsy between acetabular fracture patients whose fracture was reduced and fixated using the modified Stoppa approach (subjects) and pelvic fracture patients (controls) using physical strength testing, radiographs, clinical assessment, and a validated functional outcome questionnaire. The investigators' research hypothesis is that there will be less strength and higher incidence of obturator nerve palsy in patients treated with the modified Stoppa approach (intervention) than in patients treated without the modified Stoppa approach (controls).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the subject patient population under study consists of male and female adults, at least 18 years old, who had an acetabular fracture that was treated with the modified Stoppa approach.
* Inclusion criteria for the control patient population under study consists of male and female adults, at least 18 years old, who had acetabular fractures with similar fracture patterns as the study group that were treated with any other approach than the Stoppa approach.

Exclusion Criteria:

* Exclusion criteria for the subject and control patient population consist of:
* Patients who are non-ambulatory.
* Patients less than 18 years of age.
* Patients who do not speak English.
* Patients who are unable to complete their follow-up in Utah.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pelvic fracture patients and patients treated for acetabular fractures with the modified Stoppa approach will be asked to consent to a voluntary study investigating physical function at their 2 week follow-up appointment.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2012-04; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Outpatient physical therapy strength testing will be used to assess hip adductor strength in all participants (subjects and controls). | 1 year follow-up after surgery

SECONDARY OUTCOMES:
Radiographs and clinical assessment at follow-up appointments will be used to determine incidence of obturator nerve palsy in both groups (subjects and controls). | 1 year follow-up after surgery

CONTACTS AND LOCATIONS:
Overall Officials: David Rothberg, MD, Principal Investigator — Orthopedic Surgery Operations
Locations (1):
- University of Utah Orthopedics Center, Salt Lake City, Utah, United States